CLINICAL TRIAL: NCT03354624
Title: Cortical Neuroplasticity by Muscle Pain and Non-invasive Modulation of Pain-induced Plasticity
Brief Title: Cortical Neuroplasticity by Muscle Pain of Pain-induced Plasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Enrico De Martino, Medical Doctor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20160022
Record Dates: First submitted 2017-11-19; First posted 2017-11-28 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Nerve Growth Factor; Exercise; Motor Activity; Abnormality of SSEPs; Hyperalgesia
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Motor Activity; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nerve growth factor group (Experimental): Three injections of sterile solutions of recombinant human nerve growth factor (NGF) will be performed in the right extensor carpi radialis muscle to induce muscle hyperalgesia.
  Interventions: Drug: Sterile solutions of recombinant human nerve growth factor (NGF)
- Nerve growth factor group + delayed onset muscle soreness (Experimental): Injections of nerve growth factor and eccentric exercise of the extensor carpi radialis muscle will be performed to induce muscle hyperalgesia.
  Interventions: Drug: Sterile solutions of recombinant human nerve growth factor (NGF)

INTERVENTIONS:
Drug: Sterile solutions of recombinant human nerve growth factor (NGF) — The intramuscular injections of NGF cause muscle soreness.

SUMMARY:
The purpose of this study is to investigate the sensory-motor cortical excitability response to delayed onset muscle soreness (DOMS) on Extensor Carpi Radialis (ECR) muscle during muscle hyperalgesia provoked by nerve growth factor (NGF).

DETAILED DESCRIPTION:
The purpose of this study is to assess changes in sensory-motor cortical excitability during experimental muscle hyperalgesia across several days provoked by injections of nerve growth factor (NGF) into the Extensor Carpi Radialis (ECR) muscle and delayed onset muscle soreness (DOMS) of the ECR muscle.

It was hypothesized that muscle hyperalgesia across several days would result in:

i) Increased sensory cortical excitability, based on somatosensory evoked potentials by means of electrical stimulation of the radial nerve, (increase of central-parietal evoked-potential P45 and decrease of frontal evoked-potential N30); ii) Increased corticomotor excitability of a ECR (increase map volume and number of active sites), assessed as motor evoked potentials induced by transcranial magnetic stimulation in primary motor cortex (M1); iii) Reduction of alpha oscillation based on nociceptive stimulus-evoked suppression of alpha activity in sensory regions (recording electrodes on contra-lateral parietal area);

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Speak and understand English.

Exclusion Criteria:Pregnancy

* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* History of chronic pain or current acute pain
* Previous experience with rTMS
* Contraindications to rTMS application (history of epilepsy, metal in the head or jaw etc.).
* Failure to pass the "TASS questionnaire" (TASS = Transcranial Magnetic Stimulation Adult Safety Screen)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Pain rating | Change from baseline at 2 weeks
  Pain on an 11-point numerical rating scale (0 = no pain, 10 = most intense pain imaginable)

SECONDARY OUTCOMES:
Muscle soreness | Change from baseline at 2 weeks
  7-point Likert scale; 0 = 'a complete absence of soreness', 1 = 'a light soreness in the muscle felt only when touched/vague ache', 2 = 'a moderate soreness felt only when touched/a slight persistent ache', '3 = 'a light muscle soreness when lifting or carrying objects', 4 = 'a light muscle soreness, stiffness or weakness when moving the wrist without gripping an object', 5 = 'a moderate muscle soreness, stiffness or weakness when moving the wrist', 6 = 'a severe muscle soreness, stiffness or weakness that limits the ability to move'
Patient-rated Tennis Elbow Evaluation | Change from baseline at 2 weeks
  The Patient-rated Tennis Elbow Evaluation will be used to assess average pain and disability of the injected arm
Pressure pain thresholds | Change from baseline at 2 weeks
  Pressure applied to the surface of the skin using a handheld algometer.
Motor evoked potentials | Change from baseline at 1 week
  Transcranial magnetic stimualtion will be used to evoke motor evoked potentials (MEPs) to the extensor carpi radialis muscle
Sensory evoked potentials | Change from baseline at 1 week
  EEG recodring
Alpha oscillations | Change from baseline at 1 weeks
  Continuous EEG recording

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, North Denmark, Denmark